CLINICAL TRIAL: NCT06331611
Title: MONITORING NEUROMUSCULAR BLOCK IN PAEDIATRIC ANAESTHESIA: RANDOMISED CLINICAL STUDY
Brief Title: MONITORING NEUROMUSCULAR BLOCK IN PAEDIATRIC ANAESTHESIA
Acronym: MOTOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Nicola Disma, MD, Prof, Istituto Giannina Gaslini
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Motor
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Anesthesia,General; Neuromuscular Blockade; Tracheal Intubation
Keywords: Anesthesia; Pediatric; Neuromuscular blockade; Monitoring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TOF Monitoring (Experimental): Instrumental monitoring with electromyography (TOF Group)
  Interventions: Device: TOF monitoring
- Clinical monitoring (Standard Group) (Active Comparator): Clinical monitoring
  Interventions: Device: TOF monitoring

INTERVENTIONS:
Device: TOF monitoring — Reversal with Sugammadex will be based on TOF monitoring

SUMMARY:
To date there is still little scientific evidence regarding neuromuscular block monitoring in pediatric anesthesia and indications for safe reversal. Although the use of rocuronium and sugammadex is becoming wide, qualitative monitoring or clinical practice are applied instead of quantitative monitoring (acceleromyography-electromyography EMG). The use of neuromuscular monitoring leads to better control of intraoperative paralysis, proper timing of extubation, and reduced risk of residual postoperative paralysis-paralysis (PORC) and related complications.

The main objective of the study is to analyse the incidence of sugammadex use and the total dose/kg, with and without the aid of quantitative neuromuscular monitoring.

Secondary objectives are:

* the time required to extubate different patients,
* the incidence of respiratory complications at extubation,
* the need to administer additional doses of sugammadex. A prospective RCT. Patients will be divided into two study groups; in the first group, quantitative neuromuscular monitoring based on electromyography (EMG) will be used, while in the second group, the same monitoring will be applied but covered (blinded to the anesthetist) and the pharmacological strategy is based exclusively on the clinical practice All children aged between 2 months and 6 years, scheduled to undergo elective non-cardiac surgical procedures, lasting approximately from one to two hours(anesthesia time), with general anesthesia and tracheal intubation receiving a non-depolarizing blockade agent.
* Children between 2 months and 6 years
* Children who will undergo elective non cardiac surgery (maximum two hours of anesthesia time with tracheal intubation receiving a non depolarizing blockade agent),
* Acquisition of informed consent by a legally recognized representative capable of understanding the document and providing consent on behalf of the participant.

  * Children under 2 months of age or over 12 years of age,
  * Children with an ASA classification > 3,
  * Presence of neuromuscular disease, channelopathy, or any clinical condition that contraindicates the administration of neuromuscular muscle relaxants,
  * Confirmed or suspected allergy to sugammadex or rocuroniumt,
  * Presence of amputation or limb malformations that make placement of neuromuscular monitoring impossible,
  * Any specific contraindication to any aspect of the protocol. 12 months The randomization process will performed using numbers randomized by a computer-generated random number sequence. The randomization list will be prepared by independent statistician . The subjects will be assigned to the treatment arm in a sequence as per the randomization code provided in a closed envelope in a 1:1 ratio. The investigator will administered the treatment as per the randomization codes.

One hundred children undergo in the clinically guided group and 100 children in the neuromuscular monitoring groups with the aim to include 200 children in total.

Demographics and baseline characteristics with mean, median, standard deviation, and range (minimum, maximum) will generated for each arm. Subject disposition, including the number of subjects withdrawn or discontinued from the study, for each arm will summarized. The study will follow the CONSORT guidelines for statistical analysis and reporting. Chi squared test or Fisher's exact test and Student's t-test or Mann Whitney test will applied to categorical and continuous data, respectively, with a significance level of 5% by two-sided test. Statistical analysis was performed using SPSS software (ver. 21.0) (IBM, Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 months to 6 years of age
* Children undergoing elective non-cardiac surgery with an estimated anesthesia time of about 60 to 120 minutes
* ASA ≤ 2
* Acquisition of informed consent by a legally recognised representative able to understand the document and provide consent on behalf of the participant.

Exclusion Criteria:

* Children under 2 months or over 6 years of age
* Children with ASA classification ≥ 3
* Presence of neuromuscular diseases, channelopathies or any clinical condition contraindicating the administration of neuromuscular muscle relaxants
* Confirmed or suspected allergy to the active substance
* Presence of amputation or limb malformations that make the positioning of neuromuscular monitoring impossible
* Any specific contraindication to any aspect of the protocol

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sugammadex administration | End of anesthesia
  The primary objective will be to analyse the differences in the choice of per kilogram dosage of sugammadex and the decision to administer (yes/no) used to allow the reversal of neumuscolar block (TOFr ≥ 0.9) based on whether or not neuromuscular monitoring is used.

IPD SHARING:
Plan to Share IPD: No